# PINPOINT: Gaming Technology to Engage Adolescent Sickle Cell Patients in Precision Pain Management

**Usability Protocol** 

NCT03291613

July 2018

## PINPOINT PHASE I USABILITY PROTOCOL

#### **PROCEDURES**

Usability testing is a part of Specific Aim #5, which is to conduct a series of usability testing with 13-17-year-olds with sickle cell disease (SCD). These sessions were conducted in order to assess app functionality, navigation, and satisfaction.

Usability sessions were led by a project coordinator at Klein Buendel in Golden, CO. Each session occurred over the web using Zoom videoconferencing and were approximately 1 hour in length.

Participants were asked to complete defined tasks within the Pinpoint app, including completion of the PAT. Participants were also asked to complete either the APPT or PROMIS, and System Usability Scale (SUS) measures on paper.

The sessions were audio recorded via Zoom videoconferencing software.

Although identifiers such as name, email address, and phone number were used for the collection of the data, all identifiers are stored in secure files and behind computer firewalls and results will be shared in combined form only. Also, disclosure of participants' responses cannot reasonably be expected to place the subjects at risk of criminal or civil liability, or be damaging to their financial standing, employability, or reputation.

### RECRUITMENT

Participants were recruited from a list of previous focus group participants and Sickle Cell Disease Association of America (SCDAA) chapters located across the country. All participants (n=12) were 13-17 years old, had been diagnosed with Sickle Cell Disease, and consented to participate.

#### SCREENING

A project coordinator at KB screened the participants based on the study criteria. Participants had to be between the age of 13 and 17 years, be diagnosed with SCD, able to speak and read English, and have parental consent to participate and assent to participate.